CLINICAL TRIAL: NCT01897935
Title: Flare Photometry in Uveitis Patients
Status: Completed | Type: Observational
Sponsor: ChromoLogic, LLC (Industry)
Collaborators: UW Medicine Eye Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: OFAM_PRO_120417
Record Dates: First submitted 2013-07-08; First posted 2013-07-12 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Uveitis
Keywords: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a cross sectional study of a novel non-invasive optical flare photometer (OFAM). Patients meeting the inclusion/exclusion criteria will receive a standard eye examination including a slit lamp examination to collect ocular flare data. In addition to the standard eye examination, subjects will receive flare measurements using the OFAM device.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Ability to understand and willingness to sign a written informed consent document.
* To be eligible for the uveitis arm of the study subjects must have active anterior chamber uveitis in one or both eyes as determined by a physician
* To be eligible for the non-inflammatory arm of the study the study subjects must have no ocular inflammation in either eye as determined by a physician.

Exclusion Criteria:

* Inability to give informed consent
* Exclusion criteria for the uveitis arm: no active disease
* Exclusion criteria for the non-inflammatory arm: Signs of uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with uveitis seen in the uveitis clinic at the UW Medicine Eye Institute would be eligible for participation in the uveitis arm of the study (n ≤ 50). Patients with other, non-inflammatory forms of eye disease will be eligible for the non-inflammatory arm of the study (n ≤ 50).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Establish OFAM algorithms for quantitation of ocular flare | 3 months
  OFAM algorithms for quantitation of ocular flare will be established by comparing the output of the OFAM device to the flare measurements obtained during the standard slit lamp examination.

SECONDARY OUTCOMES:
Determine the impact that various potential confounders such as age and sex have on OFAM Measurements | 3 months
  OFAM data for various sub-groups (age and sex) will be compared in order to evaluate the degree to which each sub-group acts as a confounder for OFAM measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Lam, MD, Principal Investigator — UW Medicine Eye Institute; Russell Van Gelder, MD, Principal Investigator — UW Medicine Eye Institute
Locations (1):
- UW Medicine Eye Institute, Seattle, Washington, United States